CLINICAL TRIAL: NCT00370045
Title: Peri-Procedural Myocardial Infarction, Platelet Reactivity, Thrombin Generation, and Clot Strength: Differential Effects of Eptifibatide + Bivalirudin Versus Bivalirudin -The CLEAR PLATELETS-2 Study
Brief Title: Peri-Procedural Myocardial Infarction, Platelet Reactivity, Thrombin Generation, and Clot Strength: Differential Effects of Eptifibatide + Bivalirudin Versus Bivalirudin
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LifeBridge Health (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04745
Record Dates: First submitted 2006-08-28; First posted 2006-08-30 (Estimated); Last update posted 2006-08-30 (Estimated); Status verified 2006-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — bivalirudin; Eptifibatide

INTERVENTIONS:
Drug: Bivalirudin with and without eptifibatide

SUMMARY:
The purpose of this study is to compare levels of clot formation (platelet aggregation), markers of heart muscle damage, and inflammation in two groups undergoing percutaneous coronary stent implantation. The first group will be on a regimen of high-dose clopidogrel used in combination with bivalirudin plus eptifibatide, and the second group will be on a regimen of high-dose clopidogrel with bivalirudin alone. Clinical outcomes will be determined up to one year after enrollment.

DETAILED DESCRIPTION:
Percutaneous stent implantation has revolutionized the revascularization procedure for patients with obstructive coronary disease and angina. The major risk of coronary stenting, both during and after the procedure, is clot formation (thrombosis) which often leads to significant heart muscle damage. The standard medical practice for patients undergoing coronary stenting is the use of antiplatelet (plavix, aspirin) and anticoagulant (blood thinner) therapy. The results from our recently completed CLEAR PLATELETS I study showed that the addition of eptifibatide (a potent antiplatelet agent) to current therapy resulted in superior reduction in clot formation, inflammation and heart damage after elective coronary intervention. Recent studies have also suggested the drug bivalirudin to be a safer and more effective therapy compared to heparin, the current anticoagulant agent of choice. It has been hypothesized that bivalirudin acts not only as an anticoagulant but also as an antiplatelet agent, making the use of eptifibatide in current coronary therapy unwarranted. In the CLEAR PLATELET II study, we will compare levels of clot formation (platelet aggregation), markers of heart muscle damage, and inflammation in two groups. The first group will be on a regimen of high-dose clopidogrel used in combination with bivalirudin plus eptifibatide, and the second group will be on a regimen of high-dose clopidogrel with bivalirudin alone. The antiplatelet/antithrombotic effect that bivalirudin has in combination with these current therapies is unknown; therefore we hope to see the effect that bivalirudin has on arresting platelet formation with and without eptifibatide.

This research will be done at Sinai Hospital of Baltimore with Paul Gurbel M.D. as the principal investigator. It will include 200 patients who will be randomized equally between groups.

Clopidogrel (600 mg) + eptifibatide + bivalirudin Clopidogrel (600 mg) + bivalirudin

All patients will receive treatment with clopidogrel in the cath lab immediately after successful stenting. All patients post-stenting will receive standard antiplatelet treatment (75mg Plavix and 325 mg aspirin). Patients will have serial assessment of platelet reactivity, myocardial necrosis markers, and inflammatory markers (3 tablespoons of blood per time point) at baseline, 2 hours, 8 hours, and 18- 24 hours post-stenting. All blood work will be processed at the Sinai Center for Thrombosis Research. Clinical outcomes will be recorded using a standard case report form. Patients will be followed up at 30 days and 1 year by telephone to assess for adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Subjects (men or women) aged ³ 18
* Patients undergoing elective coronary stenting (200 patients)

Exclusion Criteria:

* ST-segment elevation myocardial infarction within 48 hours prior to randomization
* Prior PCI within previous 4 weeks of randomization or planned staged PCI within the subsequent month.
* Cardiogenic shock
* > 50% unprotected left main stenosis
* Any low molecular weight heparin within the prior 12 hours
* Treatment with any P2Y12 blocker (Plavix or Ticlid) within the previous 14 days before randomization
* Treatment with any platelet GPIIb/IIIa inhibitor within the previous 30 days before randomization
* Concurrent treatment with warfarin
* History of bleeding diathesis, or evidence of active abnormal bleeding within 30 days of randomization.
* History of hemorrhagic stroke at any time, or stroke or TIA of any etiology within 30 days of randomization.
* Major surgery within 6 weeks prior to randomization.
* Known platelet count of <100,000/mm3.
* PT > 1.5 X control
* HCT < 25%
* Known allergy or contraindication to eptifibatide, heparin, aspirin or plavix.
* Participation in a study of experimental therapy or device 30 days prior to randomization.
* Creatinine level of greater than 2.0 mg/dl or a creatinine clearance <30mL
* Known history of alcohol or drug abuse
* Pregnant women or women of child bearing potential not using an acceptable method of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2006-03

PRIMARY OUTCOMES:
Compare the antiplatelet effects of clopidogrel+bivalirudin vs. clopidogrel+bivalirudin+eptifibatide in patients undergoing elective percutaneous intervention

SECONDARY OUTCOMES:
Compare the release of myocardial necrosis and inflammatory markers
Measure platelet reactivity with conventional light transmittance aggregometry and thrombelastography
Assess in-hospital 30 day, and 1 year clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, MD, Principal Investigator — Platelet and Thrombosis Research L.L.C
Locations (1):
- Sinai Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Lewis JP, Ryan K, O'Connell JR, Horenstein RB, Damcott CM, Gibson Q, Pollin TI, Mitchell BD, Beitelshees AL, Pakzy R, Tanner K, Parsa A, Tantry US, Bliden KP, Post WS, Faraday N, Herzog W, Gong Y, Pepine CJ, Johnson JA, Gurbel PA, Shuldiner AR. Genetic variation in PEAR1 is associated with platelet aggregation and cardiovascular outcomes. Circ Cardiovasc Genet. 2013 Apr;6(2):184-92. doi: 10.1161/CIRCGENETICS.111.964627. Epub 2013 Feb 7. PMID 23392654
- [Derived] Shuldiner AR, O'Connell JR, Bliden KP, Gandhi A, Ryan K, Horenstein RB, Damcott CM, Pakyz R, Tantry US, Gibson Q, Pollin TI, Post W, Parsa A, Mitchell BD, Faraday N, Herzog W, Gurbel PA. Association of cytochrome P450 2C19 genotype with the antiplatelet effect and clinical efficacy of clopidogrel therapy. JAMA. 2009 Aug 26;302(8):849-57. doi: 10.1001/jama.2009.1232. PMID 19706858
- [Derived] Gurbel PA, Bliden KP, Saucedo JF, Suarez TA, DiChiara J, Antonino MJ, Mahla E, Singla A, Herzog WR, Bassi AK, Hennebry TA, Gesheff TB, Tantry US. Bivalirudin and clopidogrel with and without eptifibatide for elective stenting: effects on platelet function, thrombelastographic indexes, and their relation to periprocedural infarction results of the CLEAR PLATELETS-2 (Clopidogrel with Eptifibatide to Arrest the Reactivity of Platelets) study. J Am Coll Cardiol. 2009 Feb 24;53(8):648-57. doi: 10.1016/j.jacc.2008.10.045. PMID 19232896